CLINICAL TRIAL: NCT03737448
Title: A Phase 1b Open-Label Study Assessing the Pharmacokinetics, Tolerability, and Safety of Oral Trimetazidine in Subjects With Acute-on-Chronic Liver Failure
Brief Title: TRimetazidine for acUte on Chronic Liver Failure STudy
Acronym: TRUST
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Martin Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MP-0614-001
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Trimetazidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): * AD with serum creatinine ≥ 1 and < 2 mg/dL, OR
  * ACLF 1 with
    * liver failure and serum creatinine ≥ 1.5 and < 2 mg/dl, or
    * liver failure and West Haven grade 1-2 hepatic encephalopathy, or
    * coagulation failure and serum creatinine ≥ 1.5 and < 2 mg/dl, or
    * coagulation failure and West Haven grade 1-2 hepatic encephalopathy, OR
  * ACLF 2 with
    * liver failure and coagulation failure, or
    * liver failure and West Haven grade 3-4 hepatic encephalopathy.
  Interventions: Drug: Trimetazidine
- Group 2 (Experimental): * ACLF 1 with renal failure (serum creatinine ≥ 2.0 and < 3.5 mg/dL), OR
  * ACLF 2 with
    * liver failure and renal failure (serum creatinine ≥ 2.0 and < 3.5 mg/dL), or
    * coagulation failure and renal failure (serum creatinine ≥ 2.0 and < 3.5 mg/dL).
  Interventions: Drug: Trimetazidine

INTERVENTIONS:
Drug: Trimetazidine — Subjects with receive up to 60 mg daily

SUMMARY:
The study will assess the pharmacokinetics (PK), tolerability, and safety of oral trimetazidine administered to subjects with AD (ACLF Grade 0) or with ACLF Grade 1 or 2.

DETAILED DESCRIPTION:
The study will assess the PK, tolerability, and safety of oral trimetazidine administered to subjects with acute-on-chronic (ACLF) Grades 1 and 2 with liver failure and a range of renal function. Subjects will receive up to 60 mg/day for 28 days.

Two groups of subjects will be enrolled:

Group 1

* AD with serum creatinine ≥ 1 and < 2 mg/dL, OR
* ACLF 1 with

  * liver failure and serum creatinine ≥ 1.5 and < 2 mg/dl, or
  * liver failure and West Haven grade 1-2 hepatic encephalopathy, or
  * coagulation failure and serum creatinine ≥ 1.5 and < 2 mg/dl, or
  * coagulation failure and West Haven grade 1-2 hepatic encephalopathy, OR
* ACLF 2 with

  * liver failure and coagulation failure, or
  * liver failure and West Haven grade 3-4 hepatic encephalopathy.

Group 2

* ACLF 1 with renal failure (serum creatinine ≥ 2.0 and < 3.5 mg/dL), OR
* ACLF 2 with

  * liver failure and renal failure (serum creatinine ≥ 2.0 and < 3.5 mg/dL), or
  * coagulation failure and renal failure (serum creatinine ≥ 2.0 and < 3.5 mg/dL).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years, inclusive, at screening.
2. Stable diagnosis of AD, ACLF Grade 1 or ACLF Grade 2 for no less than 2 days (as determined at the discretion of the investigator)*.
3. Anticipated duration of hospital stay of at least 7 days.
4. For Group 1:

   * AD with SCr ≥ 1 and < 2 mg/dL, OR
   * ACLF 1 with

     * Tbil ≥ 12 mg/dL, SCr ≥ 1.5 and < 2 mg/dl, and HE 0-2, or
     * Tbil ≥ 12 mg/dL, and SCr < 1.5 mg/dL, and HE 1-2, or
     * INR ≥ 2.5, SCr ≥ 1.5 and < 2 mg/dl, and HE 0-2, or
     * INR ≥ 2.5, SCr < 1.5 mg/dL, and HE 1-2, OR
   * ACLF 2 with

     * Tbil ≥ 12 mg/dL, INR ≥ 2.5, and SCr < 2 mg/dL, or
     * Tbil ≥ 12 mg/dL, HE 3-4, and SCr < 2 mg/dL
5. For Group 2:

   * ACLF 1 with SCr ≥ 2.0 and < 3.5 mg/dL, OR
   * ACLF 2 with

     * Tbil ≥ 12 mg/dL, and SCr ≥ 2 and < 3.5 mg/dL, or
     * INR ≥ 2.5, and SCr ≥ 2 and < 3.5 mg/dL.
6. Female patients must be of non-childbearing potential, or, if non-sterile, must agree to sexual abstinence or use a highly effective method of contraception from Screening to 3 days after the final dose.
7. Non sterile male patients must agree to sexual abstinence or use a highly effective method of contraception from Screening to 3 days after the final dose if sexually active.
8. Able to comprehend and willing to sign an informed consent form, or, if unable to consent, consent is conducted per local requirements.

Exclusion Criteria:

1. Diagnosis of AD or ACLF (of any grade) >14 days before enrollment*.
2. Circulatory failure.
3. Respiratory failure i.e. PaO2/FiO2 ≤ 200 and/or baseline SpO2/FiO2 ≤ 214.
4. Brain failure (West Haven grade 3 or 4 hepatic encephalopathy) with coagulation failure (INR > 2.5).
5. Gastrointestinal bleeding within 72 hours prior to enrollment. (Subjects who fail this criterion may qualify after 72 hours).
6. Uncontrolled bacterial infection (urinary tract infection, spontaneous bacterial peritonitis, pneumonia, bacteremia, soft tissue infections, etc.) (as determined at the discretion of the investigator).
7. Invasive fungal infection.
8. Platelet count <30,000 cells/mL.
9. White blood cell count <1000 cells/uL.
10. Patients on hemodialysis or continuous venovenous hemofiltration.
11. Patients who have undergone or are scheduled for imminent organ transplantation. (Patients may be on a transplant list as long as no date has been set for transplantation)
12. Hospitalization for ACLF within the 3 months prior to screening.
13. History of hepatocellular carcinoma, unless within Milan Criteria (up to 3 lesions each < 3 cm or 1 lesion < 5 cm; no extrahepatic involvement; no evidence of gross vascular invasion).
14. Active non-hepatic malignancy.
15. Parkinson's disease, Parkinsonian-type symptoms (gait disorder, tremor, etc.), restless leg syndrome or other movement disorders other than asterixis.
16. Fulminant Wilson's, fulminant autoimmune hepatitis, or Budd-Chiari syndrome.
17. Septic shock (hypotension requiring vasopressors to maintain a mean arterial pressure of 65 mm Hg or greater and having a serum lactate level greater than 2 mmol/L (> 18 mg/dL) after adequate fluid resuscitation.
18. Patients who have undergone placement of a transjugular intrahepatic portosystemic shunt (TIPS) or surgical shunt in the past 6 months.
19. Any invasive procedure within 48 hours prior to enrollment with high risk of uncontrolled bleeding (as determined at the discretion of the investigator).
20. Female with a positive pregnancy test or lactating.
21. Positive results for human immunodeficiency virus HIV-1 or HIV-2.
22. Current treatment with trimetazidine.
23. Known allergy to trimetazidine or excipients.
24. Currently receiving an investigational treatment.
25. Any condition that, in the opinion of the Investigator (or designee), would limit the subject's ability to complete or participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
plasma pharmacokinetics | 28 days
  Cmax
plasma pharmacokinetics | 28 days
  AUC

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events [Safety and Tolerability] | 90 days
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Martin Pharmaceuticals
Locations (24):
- Austria (3):
  - Medical University of Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna
- Belgium (2):
  - University of Antwerp, Antwerp
  - Erasme Hospital, Brussels
- France (4):
  - Hospital Claude Huriez, Lille
  - Hospital Pitie-Salpetriere, Paris
  - Rennes University Hospital, Rennes
  - Hôpital Paul Brousse, Villejuif
- Germany (7):
  - University of Essen, Essen
  - JW Goethe Clinic, Frankfurt
  - Universitätsklinikum Halle Klinik und Poliklinik für Innere Medizin I, Halle
  - University of Hannover, Hanover
  - University of Heidelberg, Heidelberg
  - University of Leipzig, Leipzig
  - University of Münster, Münster
- Spain (8):
  - Hospital Clinic, Barcelona
  - Hospital Valle de Hebron, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Gregorio Marañón, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Marques de Valdecilla Santander, Santander
  - Hospital Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No